CLINICAL TRIAL: NCT06566768
Title: A Phase 1, Open-label, Single-dose Study to Evaluate the Pharmacokinetics of Deucravacitinib (BMS-986165) Administered as Various Solid Oral Gastro-retentive Tablet Formulation Prototypes in Healthy Participants
Brief Title: Study to Evaluate Drug Levels of Various Solid Gastro-retentive Formulations of Deucravacitinib (BMS-986165) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IM011-1201
Record Dates: First submitted 2024-08-21; First posted 2024-08-22 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Healthy Participants
Keywords: Deucravacitinib; BMS-986165; Healthy volunteers; Single-dose
MeSH Terms: interventions — deucravacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part A: Deucravacitinib (Experimental)
  Interventions: Drug: Deucravacitinib
- Part B: Deucravacitinib (Experimental)
  Interventions: Drug: Deucravacitinib

INTERVENTIONS:
Drug: Deucravacitinib — Specified dose on specified days
  Other Names: BMS-986165

SUMMARY:
The purpose of this study is to identify drug levels of gastro-retentive (GR) formulations which prolong retaining time in the stomach of deucravacitinib (BMS-986165) in Healthy Participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and healthy females according to the assessment of the Investigator.
* Body mass index of 18.0 kg/m^2 through 32.0 kg/m^2, inclusive, and body weight ≥ 50 kg.

Exclusion Criteria:

* Any significant acute or chronic medical illness.
* Current or recent (within 3 months of first dose) gastrointestinal (GI) disease that could possibly affect drug absorption, distribution, metabolism, and excretion.
* History of any significant drug allergy.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to approximately 5 days
Concentration at 24 hours post dose (C24) | Up to approximately 5 days
Area under the concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-T)] | Up to approximately 5 days

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to approximately 1 month
Incidence of serious adverse events (SAEs) | Up to approximately 1 month
Incidence of AEs leading to discontinuation | Up to approximately 1 month
Incidence of participants with vital sign abnormalities | Up to approximately 1 month
Incidence of participants with electrocardiogram (ECG) abnormalities | Up to approximately 1 month
Incidence of participants with physical examinations abnormalities | Up to approximately 1 month
Incidence of participants with clinical laboratory abnormalities | Up to approximately 1 month
Time of maximum observed concentration (Tmax) | Up to approximately 5 days
Apparent terminal plasma half-life (T-HALF) | Up to approximately 5 days
Apparent total body clearance (CLT/F) | Up to approximately 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com